CLINICAL TRIAL: NCT03004066
Title: Daptomycin Concentration in Drainage Fluid and Blood Samples of ICU Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: Dapto
Record Dates: First submitted 2016-11-16; First posted 2016-12-28 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2018-04

CONDITIONS: Heart Assist Device
MeSH Terms: interventions — Daptomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Daptomycin — standard care

SUMMARY:
10 patients with chronic heart failure receiving daptomycin therapy after implantation of a left ventricular heart assist system. Measurement of daptomycin levels in drainage fluids (mediastinal and pleural drainage systems) and in blood samples.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* heart assist device implantation
* wound drainage
* daptomycin therapy

Exclusion Criteria:

* pregnancy
* no written consent possible
* absence of wound drainage
* allergy to study medication
* acute rhabdomyolysis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients after heart assist device implantation with wound drainage receiving daptomycin therapy
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
levels of Daptomycin in drainage fluid | 4 days
  Pharmacokinetics of Daptomycin in intensive care patients with wound drainage after surgery (LVAD implantation)
levels of Daptomycin in blood samples | 4 days
  Pharmacokinetics of Daptomycin in intensive care patients after surgery (LVAD implantation)

SECONDARY OUTCOMES:
infections | 14 days
  incidence of gram-positive infections

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Prohaska, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No